CLINICAL TRIAL: NCT04027920
Title: Disastrous Delayed Postpartum Hemorrhage After Three Days of Shenghua Decoction Treatment: a Case Report
Brief Title: Postpartum Hemorrhage After Shenghua Decoction Treatment
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 108046-C
Record Dates: First submitted 2019-07-12; First posted 2019-07-22 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2019-07

CONDITIONS: Postpartum Hemorrhage
Keywords: postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Shenghua Decoction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Shenghua Decoction — Three days' shenghua decoction treatment

SUMMARY:
A rare case of disastrous delayed postpartum hemorrhage after three days of shenghua decoction treatment.

DETAILED DESCRIPTION:
A rare case of disastrous delayed postpartum hemorrhage after three days of shenghua decoction treatment.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum hemorrhage after shenghua decoction treatment.

Exclusion Criteria:

* Nil

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: A postpartum woman with delayed pospartum hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Presence of postpartum hemorrhage or not | 1 year
  Presence of postpartum hemorrhage or not, following three days of shenghua decoction treatment. The total estimated blood loss was approximately 2000 mL at that time. Her hemoglobin was revealed to be 2.6 g/dL, her hematocrit was 8.5%, and the vaginal bleeding persisted despite medications, so emergency total hysterectomy was performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided